CLINICAL TRIAL: NCT00788073
Title: A Double-Blind, Placebo-Controlled, Crossover, Flexible-Dose Evaluation of the Efficacy, Safety and Tolerability of STX209 in the Treatment of Irritability in Subjects With Fragile X Syndrome
Brief Title: Safety, Tolerability and Efficacy Study of STX209 in Subjects With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seaside Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22001
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Results first posted 2013-05-06 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-03

CONDITIONS: Fragile X Syndrome
Keywords: fragile X syndrome; irritability; behavior problems
MeSH Terms: conditions — Fragile X Syndrome; Mental Disorders | interventions — arbaclofen placarbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STX209 (Active Comparator): STX209 variable dose from 1mg bid to 10mg tid, capsule, oral, 4 weeks
  Interventions: Drug: STX209
- Placebo (Placebo Comparator): variable dose (same flexible dose titration protocol), bid to tid, capsule, Oral, 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STX209 — Variable dose from 1 mg bid to 10 mg tid, Capsule, Oral, 4 weeks
  Other Names: arbaclofen
  Arms: STX209
Drug: Placebo — variable dose (same flexible dose titration protocol), bid to tid, capsule, Oral, 4 weeks
  Arms: Placebo

SUMMARY:
The study objective is to explore the efficacy, safety and tolerability of STX209 for treatment of irritability in subjects with FSX. We hypothesize that STX209 will improve irritability and other typical problem behaviors associated with fragile X syndrome. We also hypothesize that STX209 will be safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 12 to 40 years of age eventually expanding to 6 years of age
* Molecular documentation of the fragile X mutation.
* Clinical Global Impression - Severity (CGI-S) rating for problem behavior of moderate or higher at screening and at Visit 1
* An Aberrant Behavior Checklist (ABC-C) Irritability Subscale score >12 and at least 3 items on the Irritability Subscale rated at least moderate or above.
* Current treatment with no more than three psychoactive medications, including anti-epileptics.
* Current pharmacological treatment regimen has been stable for at least 4 weeks.

Exclusion Criteria:

* Subjects with a history of seizure disorder who are not currently receiving treatment with antiepileptics.
* Subjects with any condition, including alcohol and drug abuse, which might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. This includes, but is not limited to impairment of renal function, evidence or history of malignancy or any significant hematological, endocrine, cardiovascular, respiratory, hepatic, or gastrointestinal disease.
* Subjects who plan to initiate or change pharmacologic or non-pharmacologic interventions during the course of the study.
* Subjects who are currently receiving treatment with racemic baclofen.
* Subjects currently treated with vigabatrin or tiagabine.
* Subjects taking another investigational drug currently or within the last 30 days.

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Berry-Kravis, MD, PhD, Principal Investigator — Rush University Medical Center; Randi Hagerman, MD, Principal Investigator — M.I.N.D. Institute; Craig Erikson, MD, Principal Investigator — Riley Hospital for Children; Bryan King, MD, PhD, Principal Investigator — Seattle Children's Hospital; James McCracken, MD, Principal Investigator — University of California, Los Angeles; Jonathan Picker, MBChB, PhD, Principal Investigator — Boston Children's Hospital; Linmarie Sikich, MD, Principal Investigator — University of North Carolina Neurosciences Hospital; Jeremy Veenstra-VanderWeele, MD, Principal Investigator — Vanderbilt Kennedy Center; Ted Brown, MD, PhD, Principal Investigator — NYS institute for Basic Research in Developmental Disabilities; Lawrence Ginsberg, MD, Principal Investigator — Red Oaks Psychiatry Associates, PA; Shivkumar Hatti, MD, Principal Investigator — Suburban Research Associates; Raun Melmed, MD, Principal Investigator — Southwest Autism Research & Resource Center
Locations (12):
- United States (12):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - University of California-Los Angeles Neuropsychiatric Institute, Los Angeles, California
  - M.I.N.D. Institute, Sacramento, California
  - Rush University Medical Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital Boston, Boston, Massachusetts
  - NYS Institute for Basic Research in Developmental Disabilities, Staten Island, New York
  - University of North Carolina Neurosciences Hospital, Chapel Hill, North Carolina
  - Suburban Research Associates, Media, Pennsylvania
  - Vanderbilt Kennedy Center, Nashville, Tennessee
  - Red Oaks Psychiatry Associates, P.A., Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- STX209:Placebo: First Intervention=STX209 (STX209 variable dose from 1mg bid to 10mg tid, capsule, oral) Second Intervention=Placebo (Placebo variable dose (same flexible dose titration protocol) bid to tid, oral)
  Study Design:
  Placebo-controlled, Crossover study. First Intervention(28 Days)-> Withdrawal(14 Days) -> Washout(7 Days)-> Withdrawal (14 Days) Participants received all interventions.
- Placebo:STX209: First Intervention=Placebo (Placebo variable dose (same flexible dose titration protocol) bid to tid, oral) Second Intervention=STX209 (STX209 variable dose from 1mg bid to 10mg tid, capsule, oral)
  Study Design:
  Placebo-controlled, Crossover study. First Intervention(28 Days)-> Withdrawal(14 Days) -> Washout(7 Days)-> Withdrawal (14 Days) Participants received all interventions.
Period: STX209 Then Placebo
Arm/Group | STX209:Placebo | Placebo:STX209
Started | 30 | 33
Completed | 29 | 30
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — unable to return due to travel | 0 | 1
Period: Placebo Then STX209
Arm/Group | STX209:Placebo | Placebo:STX209
Started | 29 | 30
Completed | 27 | 29
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- STX209: STX209 Variable dose, 1mg bid to 10mg tid, oral capsules, 4weeks
- Placebo: placebo variable dose (same flexible dose titration protocol) bid to tid, oral, 4weeks
- Total: Total of all reporting groups
Arm/Group | STX209 | Placebo | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 24 | 46
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 14.2 (7.29) | 13.9 (6.39) | 14.1 (6.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 28 | 27 | 55
Region of Enrollment [Number; unit: participants]
  United States | 30 | 33 | 63

OUTCOME MEASURES:

1. Primary Outcome: Aberrant Behavior Checklist Irritability Subscore
Description: The Aberrant Behavior Checklist-Community Edition (ABC-C) is a 58-item questionnaire composed of five different independent subscales. The questionnaire is completed by the parent/caregiver and lists aberrant behaviors and asks about the severity of the problem. ABC-Irritability is one of the subscales and comprises of 15 items. Minimum score is 0, maximum is 45. A decreased score indicates few aberrant behaviors and clinical improvement. The entire ABC-C assessment is administered at baseline and then at the end of each Intervention Period (4 weeks after Baseline).
Time Frame: After 4 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Arm/Group | STX209:Placebo | Placebo:STX209
Number analyzed (Participants) | 63 | 63
Points on a scale | -5.1 (0.95) | -5.3 (0.95)
Statistical Analysis 1: Comparison: STX209:Placebo vs Placebo:STX209; Test type: Superiority or Other; p = 0.05, ANCOVA; Mean Difference (Final Values) = -0.2

2. Post Hoc Outcome: ABC-FXS Social Avoidance Subscore
Description: After completion of the study, but during data analysis, the ABC-C assessment was independently re-validated in Fragile X Syndrome subjects. The subscales were re-factored into a Fragile-X Syndrome specific ABC-C (ABC-FX). The ABC-FX contains the same 58 questions as the original ABC-C but there are six subscales. One of the subscales is Social Avoidance, which consists of 4 items. Minimum score is 0, maximum is 12. A decreased score indicates fewer social avoidant behaviors. A post-hoc analysis was performed from the study data examining the social avoidance subscale of the ABC-FX.
Time Frame: 4 week treatment period
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Arm/Group | STX209:Placebo | Placebo:STX209
Number analyzed (Participants) | 63 | 63
Points on a scale | -1.2 (0.24) | -0.1 (0.24)
Statistical Analysis 1: Comparison: STX209:Placebo vs Placebo:STX209; Test type: Superiority or Other; p = 0.008, ANCOVA; Mean Difference (Final Values) = 1.0

ADVERSE EVENTS:
Arm/Group | STX209 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/63
Other Adverse Events (participants affected / at risk) | 42/63 | 31/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STX209 (N=63) | Placebo (N=63)
increased irritability (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STX209 (N=63) | Placebo (N=63)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6)
headache (Nervous system disorders) | 5 (5) | 1 (1)
sedation (Nervous system disorders) | 5 (5) | 1 (1)
fatigue (General disorders) | 4 (4) | 1 (1)
irritability (Psychiatric disorders) | 4 (4) | 4 (4)
diarrhea (Gastrointestinal disorders) | 3 (3) | 5 (5)
increased appetite (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
aggression (Psychiatric disorders) | 3 (3) | 4 (4)
nasopharyngitis (Infections and infestations) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Seaside Therapeutics agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.